CLINICAL TRIAL: NCT00977795
Title: A Phase 1 and 2 Study of 5-aminolevulinic Acid (5-ALA) to Enhance Visualisation and Resection of Malignant Glial Tumors of the Brain
Brief Title: A Study of the Specificity and Sensitivity of 5-ALA Fluorescence in Malignant Brain Tumors
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI moving to Southern Illinois University to start new protocol
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EH09-377
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Brain Neoplasms
Keywords: Brain Neoplasms; 5-ALA; Aminolevulinic acid; Fluorescence; Gliomas; Glioblastoma; Surgery
MeSH Terms: conditions — Brain Neoplasms; Glioma; Glioblastoma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tumor fluorescence (Experimental): A single arm in this open-label study where all patients are treated with the study drug. Areas of the brain that are fluorescent and areas that are not fluorescent are evaluated for presence of tumor cells
  Interventions: Drug: 5-aminolevulinic acid

INTERVENTIONS:
Drug: 5-aminolevulinic acid — oral doses in phase 1 study of 10mg/kg, 20 mg/kg, 30 mg/kg, 40 mg/kg and 50 mg/kg
  Other Names: 5-ALA; aminolevulinic acid

SUMMARY:
Extent of resection is a very important prognostic factor affecting survival in individuals diagnosed with a malignant glioma. However, the infiltrative nature of the malignant glioma tumor cells produces indistinct borders between normal and malignant tissues, and the lack of easily identifiable tumor margins confounds attempts at total resection. The investigators propose to identify the borders of malignant gliomas intraoperatively using oral 5-aminolevulinic Acid (5-ALA) which results in fluorescence of the malignant cells and thereby provide an opportunity for more complete tumor resection.

When exogenous 5-ALA is provided at increased concentration the tumor cells will become fluorescent under ultraviolet light. This feature identifies the tumor cells intraoperatively and facilitates complete resection.

The following data will be collected:

* Dose-limiting toxicity data
* Tumor fluorescence assessed by neurosurgeon (0 to +++) in three distinct areas of fluorescence (Strong fluorescence, Weak fluorescence, No fluorescence)
* Tumor density from biopsies obtained by the neurosurgeon in the same three distinct areas of fluorescence and assessed by neuropathology (Solid tumor, Tumor mixed infiltrating normal brain, No tumor)
* Neurosurgeon's intra-operative estimate of residual tumor
* Neuroradiologist's estimate of post-operative residual tumor on MRI
* Time to progression by MRI
* Survival (time to progression, one year survival rate and total survival

This trial will evaluate:

* The toxicity of a single dose of oral 5-ALA given pre-operatively.
* The sensitivity and specificity of 5-ALA - Protoporphyrin IX (Pp IX) as an intraoperative fluorescent detection agent and aid for resection of tumor tissue remaining in the walls of the resection cavity of primary and recurrent malignant brain tumors.
* The relationship of the neurosurgeon's estimate of the extent of malignant glioma resection (as guided by tumor fluorescence) to the actual extent of resection determined by post-operative imaging.
* The time-to-progression, one year survival rate and total survival as a function of the extent of resection.

Following completion of the phase 1 portion of this trial, an additional 15 subjects will be entered at the recommended phase 2 dose level in order to further define the above parameters at the recommended phase 2 dose level.

DETAILED DESCRIPTION:
Specific Aims:

This study is intended to investigate the utility, safety and efficacy of 5-aminolevulinic acid (5-ALA) induced brain tumor fluorescence during malignant brain tumor resection. Specifically this study is intended to:

* Establish a safe dose for oral 5-ALA administration.
* Determine the sensitivity and specificity of 5-ALA mediated fluorescence for malignant glioma tissue in the brain.
* Compare the neurosurgeon's intra-operative estimate of the extent of malignant glioma resection (as guided by tumor fluorescence) with the actual extent of resection determined by post-operative imaging.
* Compare time-to-progression and survival to that in comparable cases performed without the aid of 5-ALA.

Background and Significance:

There is a considerable body of literature that suggests that completeness of resection is a positive factor for longer term survival in individuals with malignant glioma. Unfortunately, it is often difficult to completely remove a malignant brain tumor because during surgery it is sometimes very difficult to distinguish tumor from normal brain. It would be very helpful if there would be some way to help the surgeon make this distinction. Malignant glioma tumor cells (more so than normal cells) contain the biosynthetic pathways to produce protoporphyrin from a naturally occurring amino acid, 5-aminolevulinic acid (5-ALA). Protoporphyrin is the immediate precursor to hemoglobin (it is hemoglobin without the iron atom) and is fluorescent under blue light. When exogenous 5-ALA is provided at increased concentration, protoporphyrin concentration in the malignant cell increases at a rate far greater than normal brain cells and renders the malignant cell fluorescent red under blue light. This feature distinguishes the tumor cells from normal cells intraoperatively and facilitates complete resection.

Recent studies in Germany have confirmed the utility of pre-operative oral 5-ALA and intraoperative brain tumor fluorescence in aiding the resection of brain tumors in individuals with malignant brain tumors. These studies have led to oral 5-ALA to be approved for this indication by the European Medicines Agency (The European Medicines Agency comments and approval can be found at: http://www.emea.europa.eu/humandocs/PDFs/EPAR/gliolan/H-744-en6.pdf), but oral 5-ALA has not been approved for this indication by the United States FDA. This proposal is a phase 1 and phase 2 trial that will hopefully lead to FDA approval of oral 5-ALA for intra-operative visualization of malignant brain tumors.

Experimental Plan and Methods:

In the phase 1 part of this proposed study, a minimum of 3 to a maximum of 18 patients will be administered oral 5-ALA 4 hours prior to surgery in cohorts of 3 at five escalating doses of 5-ALA (10, 20, 30, 40, or 50 mg/kg).

The following data will be collected:

* Dose-limiting toxicity data.
* Tumor fluorescence assessed by neurosurgeon (0 to +++) in three distinct areas of fluorescence (Strong fluorescence, Weak fluorescence, No fluorescence).
* Tumor density from biopsies obtained by the neurosurgeon in the same three distinct areas of fluorescence and assessed by neuropathology (Solid tumor, Tumor mixed infiltrating normal brain, No tumor).
* Neurosurgeon's intra-operative estimate of residual tumor.
* Neuroradiologist's estimate of post-operative residual tumor on MRI.
* Time to progression by MRI.
* Survival (time to progression, one year survival rate and total survival.

This trial will evaluate:

* The toxicity of a single dose of oral 5-ALA given pre-operatively.
* The sensitivity and specificity of 5-ALA - Protoporphyrin IX (Pp IX) as an intraoperative fluorescent detection agent and aid for resection of tumor tissue remaining in the walls of the resection cavity of primary and recurrent malignant brain tumors.
* The relationship of the neurosurgeon's estimate of the extent of malignant glioma resection (as guided by tumor fluorescence) to the actual extent of resection determined by post-operative imaging.
* The time-to-progression, one year survival rate and total survival as a function of the extent of resection.

Following completion of the phase 1 portion of this trial, an additional 15 subjects will be entered at the recommended phase 2 dose level in order to further define the above parameters at the recommended phase 2 dose level.

Discussions statisticians have led to the development of a number of 2x2 tables and 3x3 tables of data analysis that will lead to establishment of the sensitivity and specificity of fluorescence-guided brain tumor resection compared to conventional brain tumor resection techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have clinically documented primary brain tumor for which resection is clinically indicated. The anticipated histology at resection should include: Anaplastic astrocytoma (10002224), Astrocytoma malignant NOS (10003572), Brain stem glioma (10006143), Ependymoma (10014967), Ependymoma malignant (10014968), Glioblastoma (10018336), Glioblastoma multiforme (10018337), Gliosarcoma (10018340), Anaplastic oligodendroglioma (10026659), Oligodendroglioma (10030286), Medulloblastoma (10027107), Mixed astrocytoma-ependymoma (10027743), Miscellaneous CNS primary tumor (10007959), Supratentorial primitive neuroectodermal tumor (10056672)
* Prior therapy is not a consideration in protocol entry
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of 5-ALA in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric phase 1 single-agent trials
* ECOG performance status <2 (Karnofsky >60%)
* Life expectancy is not a consideration for protocol entry
* Patients must have normal organ and marrow function as defined below:

  * Leukocytes > 3,000/mcL
  * Absolute neutrophil count > 1,500/mcL
  * Platelets > 100,000/mcL
  * Total bilirubin within normal institutional limits
  * AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal
  * Creatinine within normal institutional limits, OR
  * Creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* The effects of 5-ALA on the developing human fetus are unknown. 5-ALA has unknown teratogenic or abortifacient effects. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior therapy is not an exclusion criterion
* Patients may not be receiving any other investigational agents at the time of entry into the study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 5-ALA
* Personal or family history of porphyrias
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because 5-ALA is of unknown teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with 5-ALA, breastfeeding should be discontinued if the mother is treated with 5-ALA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Establish a safe dose for oral 5-ALA administration. | 6 months

SECONDARY OUTCOMES:
Determine the sensitivity and specificity of 5-ALA mediated fluorescence for malignant glioma tissue in the brain | 24 months
Compare the neurosurgeon's intra-operative estimate of the extent of malignant glioma resection (as guided by tumor fluorescence) with the actual extent of resection determined by post-operative imaging | 24 months
Compare time-to-progression and survival to that in comparable cases performed without the aid of 5-ALA | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W. Cozzens, M.D., Principal Investigator — Endeavor Health

REFERENCES:
- [Background] Keles GE, Anderson B, Berger MS. The effect of extent of resection on time to tumor progression and survival in patients with glioblastoma multiforme of the cerebral hemisphere. Surg Neurol. 1999 Oct;52(4):371-9. doi: 10.1016/s0090-3019(99)00103-2. PMID 10555843
- [Background] Sanai N, Berger MS. Glioma extent of resection and its impact on patient outcome. Neurosurgery. 2008 Apr;62(4):753-64; discussion 264-6. doi: 10.1227/01.neu.0000318159.21731.cf. PMID 18496181
- [Background] Stummer W, Pichlmeier U, Meinel T, Wiestler OD, Zanella F, Reulen HJ; ALA-Glioma Study Group. Fluorescence-guided surgery with 5-aminolevulinic acid for resection of malignant glioma: a randomised controlled multicentre phase III trial. Lancet Oncol. 2006 May;7(5):392-401. doi: 10.1016/S1470-2045(06)70665-9. PMID 16648043
- [Background] Tonn JC, Stummer W. Fluorescence-guided resection of malignant gliomas using 5-aminolevulinic acid: practical use, risks, and pitfalls. Clin Neurosurg. 2008;55:20-6. No abstract available. PMID 19248665